CLINICAL TRIAL: NCT01668381
Title: Enumeration and Function Analysis of Treg Cells in Peripheral Blood of HCC Patients Before and After Ablation Therapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Guangdong Province, Department of Science and Technology (Other Government)
Responsible Party: Principal Investigator, Ming Kuang,MD,PhD, MD,PhD, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 2010B031600209
Record Dates: First submitted 2012-03-18; First posted 2012-08-20 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; Catheter Ablation; T-Lymphocytes, Regulatory; IL-10; TGF-β; IFN-γ
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCC patients: Hepatocellular carcinoma patients treated by radiofrequency ablation
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: radiofrequency ablation — the patients are prepared by local anesthesia and intravenous sedative.guided by the ultrasound,the antenna used for radiofrequency ablation ablation is placed in the tumor to destroy tumor tissues,the output power and duration are depended by the tumor volume and location.

SUMMARY:
The purpose of this study is to determine the enumeration and function changes of regulatory t cells in peripheral blood of hepatocellular carcinoma patients before and 1 week, 4 weeks after ablation therapy.

DETAILED DESCRIPTION:
Regulatory T cells，which are also called Treg cells，play an important role in suppressing anti-tumor immunity.Accumulated evidences indicate that Treg cells are elevated in peripheral blood,however,there are also reports that decreased Treg cells are found in hepatocellular patients.This study focuses on the changes of Treg cells ratio in peripheral blood of hepatocellular carcinoma patients before and 1 week, 4 weeks after ablation ,also its functional cytokines,such as TGF-β,IL-10,IFN-γ,and inhibition function when co-cultured with CD4+CD25-、CD8+ cells. The investigators speculate that a decreased Treg ratio will be found in patients who receive ablation therapy,and its function cytokines,moreover,CD4+CD25-、CD8+ cells' proliferation and function could be inhibited when co-cultured with Treg cells.

ELIGIBILITY:
Inclusion Criteria:

* hepatocellular patients diagnosed through biopsy;or either dynamic imagine with a diagnosis of hepatocellular carcinoma and alphafetoprotein>400μg/L；or two or more dynamic imagine with a diagnosis of hepatocellular carcinoma
* Child-Pugh A or B
* well preserved renal and hematopoietic Function
* receive ablation therapy through percutaneous radiofrequency ablation or microwave ablation or ethanol injection ablation or any kind of combination of them.
* achieve complete ablation accessed by contrast-enhanced CT

Exclusion Criteria:

* incomplete ablation
* remote metastasis
* Child-Pugh C
* general infection
* autoimmune diseases
* suffer from other tumors concurrently or in last five years
* patients with immune deficit or infected by HIV
* receiving glucocorticoid or other medicine inhibiting immune system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hepatocellular carcinoma patients underwent radiofrequency ablation therapy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
variation of absolute counting of T cell subsets in peripheral blood of HCC patients before and 1,4 weeks after radiofrequency ablation therapy | 4 weeks post therapy
  changes of absolute counting of T cell subsets in peripheral blood of HCC patients before and 1,4 weeks after radiofrequency ablation therapy,such as CD3+,CD4+,CD8+,CD4+CD25+FOXP3+(Treg) cells.
variation of serum IL-10,TGF-β1,IFN-γ concentration of HCC patients before and 1,4 weeks after radiofrequency ablation therapy | 4 weeks post therapy
  variation of serum IL-10,TGF-β1,IFN-γ concentration of HCC patients before and 1,4 weeks after radiofrequency ablation therapy

SECONDARY OUTCOMES:
variation of proliferation suppression ability of CD4+CD25+ T cells of HCC patients before and 1,4 weeks after radiofrequency ablation therapy | 4 weeks post therapy
  CD4+CD25+ T cells, derived from peripheral blood of HCC patients before and 1,4 weeks after radiofrequency ablation therapy,were co-cultured with CD4+CD25- or CD8+ T cells,which were stimulated by CD3/CD28 MACSiBead Particles.CD4+CD25- and CD8+ T cells proliferation changes were analysed to test CD4+CD25+ T cell suppression ability.
variation of suppression ability of CD4+CD25+ T cells of HCC patients on cytokine secretion before and 1,4 weeks after radiofrequency ablation therapy | 4 weeks post therapy
  CD4+CD25+ T cells, derived from peripheral blood of HCC patients before and 1,4 weeks after radiofrequency ablation therapy,were co-cultured with CD4+CD25- or CD8+ T cells,which were stimulated by CD3/CD28 MACSiBead Particles.supernatant IFN-γ were analysed to test CD4+CD25+ T cell suppression ability.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, MD,PhD, Study Chair — First Affiliated Hospital, Sun Yat-Sen University; Qing-qi Ren, Bachelor, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen University,First Affiliated Hospital, Guangzhou, Guangdong, China